CLINICAL TRIAL: NCT05967975
Title: The Role of Sonoelastography in Evaluation of Therapeutic Response in Patients With Lymphoma.
Brief Title: Elastography and Treatment of Lymphoma
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Kerols Refaat Ayoub, Resident doctor, Assiut University
Other Study IDs: Elastography and lymphoma
Record Dates: First submitted 2023-07-23; First posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Elastography; Lymphoma
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To determine accuracy of elastography in assessment of superficial lymph nodes response to treatment in cases of lymphoma.

DETAILED DESCRIPTION:
Lymphomas are a heterogeneous group of malignancies that arise from the clonal proliferation of lymphocytes. It represents approximately 5% of malignancies. Overall survival is estimated to be 72%. (1)

Lymphomas are broadly classified into Hodgkin lymphoma (HL) (10%) and Non-Hodgkin lymphoma (NHL) (90%).

HL is further classified into classical and non-classical types and NHL into B-cell, T-cell and natural killer (NK) cell types. Diagnosis of lymphoma is confirmed by histopathology (FNAC, True-cut or excisional biopsy).(2) The standard treatment of lymphoma is chemotherapy and radiotherapy.

The modalities used for staging and follow up of lymphoma are:

* Computed Tomography (CT) chest, abdomen and pelvis.
* Positron Emission Tomography (PET/CT).
* Whole body Magnetic Resonance Imaging (MRI).(3)

Sonoelastography is a new technique that depends on the elastic properties of soft tissues, with the idea of malignant lesions being stiffer than benign or normal tissue. It may have a dependable role in evaluation of therapeutic response in patients with lymphoma and can be used for follow up, the same way it has been used in different parts of the body, such as the breast, and thyroid. To the best of our knowledge, there are few studies concerning the role of elastography in the field of lymphoma disease.(4)

ELIGIBILITY:
Inclusion Criteria:

* patients who are histopathologically proven as lymphoma, not receive treatment and have superficial lymphadenopathy.

Exclusion Criteria:

* 1-Lymphoma without superficial lymph nodes. 2-patients under treatment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed as lymphoma , have superficial lymph nodes and not received any treatment
Sampling Method: Probability Sample
Enrollment: 44 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
To determine accuracy of elastography in assessment of superficial lymph nodes response to treatment in cases of lymphoma. | Average three years
  Sonoelastography is a new technique that depends on the elastic properties of soft tissues, with the idea of malignant lesions being stiffer than benign or normal tissue. It may have a dependable role in evaluation of therapeutic response in patients with lymphoma and can be used for follow up, the same way it has been used in different parts of the body, such as the breast, and thyroid. To the best of our knowledge, there are few studies concerning the role of elastography in the field of lymphoma disease.

CONTACTS AND LOCATIONS:
Overall Officials: Kerols Refaat, Resident, Principal Investigator — Assiut University; Nagham Nabil, Professor, Study Director — Assiut University; Abdel-Monem Sayed, Lecture, Study Director — Assiut University